CLINICAL TRIAL: NCT01845038
Title: A Prospective, Multicenter, Randomized, Double-Masked, Multi-Arm Feasibility Study Evaluating the Safety and Efficacy of OTX-TP Compared to Timolol Drops in the Treatment of Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Multi-Arm Feasibility Study Evaluating OTX-TP Compared to Timolol in Treatment of Subjects With Open Angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTX-12-003
Record Dates: First submitted 2013-04-18; First posted 2013-05-03 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OTX-TPa (Experimental): OTX-TPa is a hydrogel punctum plug eluting travoprost in sustained release of ~4µg/day over approximately 2 months. For study masking purposes, subjects in this arm will also have natural tears drops administered.
  Interventions: Drug: OTX-TPa ~4µg/day over 2 mos. with natural tears drops
- OTX-TPb (Experimental): OTX-TPb is a hydrogel punctum plug eluting travoprost in sustained release of ~3µg/day over approximately 3 months. For study masking purposes, subjects in this arm will also have natural tears drops administered.
  Interventions: Drug: OTX-TPb ~3µg/day over 3 months with natural tears drops
- Timolol (Active Comparator): Timolol Maleate (0.5%) ophthalmic solution dosed twice daily (BID). For study masking purposes, subjects in this arm will also have a hydrogel punctum plug with no drug placed for approximately 3 months.
  Interventions: Drug: Timolol Maleate (0.5%) dosed twice daily with punctum plug without drug

INTERVENTIONS:
Drug: OTX-TPa ~4µg/day over 2 mos. with natural tears drops — OTX-TPa is a hydrogel punctum plug eluting travoprost in a sustained release of ~4µg/day over 2 months. Subjects in this arm will also receive natural tears drops.
  Arms: OTX-TPa
Drug: OTX-TPb ~3µg/day over 3 months with natural tears drops — OTX-TPb is a hydrogel punctum plug eluting travoprost in a sustained release of ~3µg/day over 3 months. Subjects in this arm will also receive natural tears drops.
  Arms: OTX-TPb
Drug: Timolol Maleate (0.5%) dosed twice daily with punctum plug without drug — Timolol Maleate (0.5%) ophthalmic solution dosed twice daily. Subjects in this arm will also have a hydrogel punctum plug without drug placed.
  Arms: Timolol

SUMMARY:
The purpose of this study is to evaluate how OTX-TP, a sustained release travoprost drug product, when placed in the canaliculus of the eyelid compares to timolol drops for the lowering of intraocular pressure (IOP) in patients with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be greater than or equal to 18 years of age at Screening.
* Subject must have a documented diagnosis of ocular hypertension, open angle glaucoma.
* Subject has a mean baseline (Day -7 and Day 0) Hour 0 (T0) untreated IOP of ≥ 24 mm Hg and ≤ 34 mm Hg in each eye, and (T0 + 4h) and (T0 + 8h) IOP of ≥ 22 mm Hg at Baseline Visit 2. Untreated IOP must be ≤ 34 mm Hg in each eye at all time points at both baseline visits.
* Subject has a BCVA of 0.6 logMAR (20/80 Snellen) or better in each eye as measured using an ETDRS chart.

Exclusion Criteria:

* Presence of any uncontrolled systemic or debilitating disease (e.g. cardiovascular disease, hypertension, diabetes, or cystic fibrosis).
* Punctum size is smaller than 0.4mm or greater than or equal to 1.0mm.
* Any single IOP in either eye at any time point during the Screening or either Baseline (Day -7/Day 0) Visits of >34 mm Hg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mean IOP change from baseline | 90 days

SECONDARY OUTCOMES:
Visualization of OTX-TP punctum plug by subject | 90 days
  OTX-TP punctum plug contains conjugated fluorescein to serve as a visualization aid through use of a blue light source and yellow filter to confirm product presence daily by subject for 90 days.

OTHER OUTCOMES:
Best corrected visual acuity | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Umhlanga Hospital Medical Centre, Durban, South Africa